CLINICAL TRIAL: NCT06975917
Title: Adjuvant Chemotherapy Regimens in Resected Biliary Tract Cancers (TOG/GI-SAFRADJU-2501)
Acronym: TOG-SAFRADJU
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Turkish Oncology Group (Network)
Responsible Party: Principal Investigator, Erman Akkus, Principle Investigator, Ankara University
Other Study IDs: i09-714-24
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Biliary Tract Cancer; Biliary Tract Cancers (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Drug Therapy; Capecitabine; Gemcitabine; gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with biliary tract cancer: Patients with biliary tract cancer, who underwent resection and received adjuvant chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Any chemotherapy regimen that is used in the adjuvant setting
  Other Names: capecitabine; gemcitabine; gemcitabine-cisplatin; gemcitabine-capecitabine; gemcitabine-oxaliplatin

SUMMARY:
The goal of this observational study is to compare chemotherapy types that are given after surgery for biliary tract cancers. The main question it aims to answer is:

Are any of the chemotherapy regimens more effective in preventing recurrence, providing longer survival, or having less toxicity?

Nationwide multicenter retrospective data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed biliary tract cancer (intrahepatic, perihilar, distal, gallbladder)
* Underwent curative-intent resection

Exclusion Criteria:

* Patients with a disease without histological confirmation
* Ampullary cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in any hospital (public, private, university/academic) across Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | From the date of adjuvant chemotherapy initiation until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 180 months
  The length of time from the start of adjuvant chemotherapy to the date of the first loco-regional or systemic recurrence or death
Overall survival | From the date of adjuvant chemotherapy initiation until the date of death from any cause, assessed up to 180 months
  The length of time from the start of adjuvant chemotherapy to the date of death

SECONDARY OUTCOMES:
2-year recurrence-free survival | From start of adjuvant chemotherapy to the date of recurrence or death in the first 2 years
  The length of time from the start of adjuvant chemotherapy to the date of recurrence or date in the first 2-years
2-year overall survival | From start of adjuvant chemotherapy to the date of death in the first 2 years
  The length of time from the start of adjuvant chemotherapy to the date of death in the first 2 years
The number of patients experienced toxicities | From the date of initiation of the first cycle of adjuvant chemotherapy until 1 month after the last cycle of adjuvant chemotherapy
  The rates of grade 1-2 and grade 3-4 toxicities, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

OTHER OUTCOMES:
Recurrence-free survival analyses in subgroups | From the date of adjuvant chemotherapy initiation until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 180 months
  Recurrence-free survival (The length of time from start of adjuvant chemotherapy to the date of the first loco-regional or systemic recurrence or death) will be analysed and compared in different subgroups.
  Subgroups
  * Age ( below 65 vs. 65 and above 65)
  * ECOG performance score (0 vs. 1)
  * Lymph node status (Positive vs negative)
  * Resection (R1 vs. R0)
  * Anatomical subtype (intrahepatic vs perihilar vs. distal vs gallbladder)
Overall survival analyses in subgroups | From the date of adjuvant chemotherapy initiation until the date of death from any cause, assessed up to 180 months
  Overall survival (The length of time from the start of adjuvant chemotherapy to the date of death) will be analysed and compared in different subgroups.
  Subgroups
  * Age ( below 65 vs. 65 and above 65)
  * ECOG performance score (0 vs. 1)
  * Lymph node status (Positive vs negative)
  * Resection (R1 vs. R0)
  * Anatomical subtype (intrahepatic vs perihilar vs. distal vs gallbladder)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine Department of Medical Oncology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.ejca.2025.115342